CLINICAL TRIAL: NCT05352438
Title: Investigation of the Effectiveness of Manual Therapy and Splint Therapy in Patients With Myofascial Temporomandibular Dysfunction Combined With Bruxism
Brief Title: Manual Therapy and Splint Therapy in Patients With Temporomandibular Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turkoglu Dr. Kemal Beyazit State Hospital (Other)
Responsible Party: Principal Investigator, Süreyya DAMAR ÖRENLER, Principal Investigator, Turkoglu Dr. Kemal Beyazit State Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-67
Record Dates: First submitted 2022-04-18; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Temporomandibular Disorder; Myofascial Pain; Bruxism
Keywords: Temporomandibular Dysfunction; Bruxism; Manual Therapy; Splint
MeSH Terms: conditions — Temporomandibular Joint Disorders; Bruxism

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy Group (Experimental): Manual Therapy combined with education and home exercises
  Interventions: Other: Manual Therapy Group
- Splint Therapy Group (Experimental): Splint Therapy combined with education and home exercises
  Interventions: Other: Splint Therapy Group

INTERVENTIONS:
Other: Manual Therapy Group — Patient education directed at parafunctional behaviors was given, and an exercise program was taught, with all the patients instructed to perform these exercises at home. The home exercise program included diaphragmatic breathing exercises, chin-tuck exercises, mandibular resistance exercises, and neck muscle stretching exercises. The patients were instructed to perform the exercises as 3 sets of 10 repetitions per day.
  In addition to the patient education and home exercises, the Manual Therapy group received a manual therapy program applied as 2 sessions of 45 mins each week for 4 weeks (total 8 sessions) by an investigator. Soft tissue and joint mobilizations were applied to the TMJ and surrounding structures and to cervical segments, trigger point treatment was applied to trigger points, and myofascial loosening was performed. Patients were instructed to perform the exercises learned in the home exercise program in 3 sets of 10 repetitions every day.
  Arms: Manual Therapy Group
Other: Splint Therapy Group — Patient education directed at parafunctional behaviors was given, and an exercise program was taught, with all the patients instructed to perform these exercises at home. The home exercise program included diaphragmatic breathing exercises, chin-tuck exercises, mandibular resistance exercises, and neck muscle stretching exercises. The patients were instructed to perform the exercises as 3 sets of 10 repetitions per day.
  In addition to the patient education and home exercises, the Splint Therapy group was given a static occlusal splint, and adjustments were made as necessary. All the patients in this group were instructed to use the splint when sleeping for a period of one month.
  Arms: Splint Therapy Group

SUMMARY:
The aim of this study was to compare the efficacy of splint treatment and manual therapy in patients diagnosed with myofascial temporomandibular dysfunction with bruxism.

DETAILED DESCRIPTION:
A total of 56 patients were evaluated. Among those, 20 patients who did not meet the criteria were excluded. 36 patients met the inclusion criteria and were willing to participate in the study.

The patients were randomly separated into two groups using the method of single- and double-digit numbers written on paper in a sealed envelope.

Those who selected a double-digit number were assigned to the manual therapy (MT) group (n:18) and those with a single-digit number to the splint therapy (ST) group (n:18).

After the further exclusion of 7 patients during the treatment period, the final evaluations were compared of 29 patients (15 MT and 14 ST) who completed the 4-week treatment process.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 50 years old,
* Patients with a diagnosis of myofascial TMD with Bruxism according to the diagnostic criteria for temporomandibular disorders (DC/TMD),
* Having pain severity ≥3 according to the Visual analogue scale (VAS),
* Probable sleep bruxism according to clinical evaluation and a questionnaire-based assessment.

Exclusion Criteria:

* Patients with a diagnosis other than myofascial TMD according to the research DC/TMD,
* a history of surgery associated with cervical and/or TMJ problems,
* a proven specific pathological condition such as cervical and/or TMJ malignancy, fracture, or systemic rheumatoid disease,
* a history of facial paralysis, a diagnosed psychiatric disease,
* if they were undergoing orthodontic treatment,
* had received physiotherapy within the last 3 months,
* or could not be co-operative.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Pain severity at 4 weeks | Baseline, 4 weeks
  Pain severity was measured with a Visual Analogue Scale (VAS), marked from 0 to 10, where 0 indicates no pain and 10 indicates intolerable pain. The patients were instructed to mark the scale corresponding to the severity of pain felt.
Change frim Baseline in Fatigue severity at 4 weeks | Baseline, 4 weeks
  Fatigue level was measured with the Fatigue Severity Scale, where patients were asked to indicate their levels of agreement with a 0-7 scale indicating "0" strong disagreement and "7" strong agreement at a total of 9 questions. A sum of all responses was calculated for analysis. Sixty-three was the maximum score. The higher value represented a higher level of fatigue.
Change from Baseline in Sleep quality at 4 weeks | Baseline, 4 weeks
  The sleep quality of patients was analyzed with the Pittsburgh Sleep Quality Index (PSQI). The PSQI includes 24 items related to both daytime and nocturnal sleep. The responses were scored from 0-3, as 7 subscores to give a global score of total points in the range of 0-21. A score of ≥5 indicated poor sleep quality.
Change from Baseline in Jaw Function limitation at 4 weeks | Baseline, 4 weeks
  Jaw function limitation was measured by the Jaw Functional Limitation Scale-20 (JFLS-20) where the patients asked for from 1 to 10 points per item (higher scores indicate worse jaw function). The JFLS-20 has 3 subscales: Mastication (6 items), Vertical Jaw Mobility (4 items), and Emotional and Verbal Expression (10 items).
Change from Baseline in Neck Disability at 4 weeks | Baseline, 4 weeks
  Neck Disability Index, consists of 10 items. Individuals included in the study were asked to give a score between 0 (no disability) and 5 (complete disability) for each item. The total score varies between 0 (no disability) and 50 (complete disability).
Change from Baseline in Patient Satisfaction questionnaire at 4 weeks. | Baseline, 4 weeks
  The Patient Satisfaction questionnaire was used to assess the patient's satisfaction with the treatment received. The patient satisfaction questionnaire (PSQ) contains 18 items tapping each of the seven dimensions of satisfaction with medical care measured by the PSQ-18.
Change from Baseline in Headache severity at 4 weeks | Baseline, 4 weeks
  The Headache Impact Test-6 (HIT-6) was used to assess the headache. The 6-item scale evaluates the frequency, the degree of restriction to daily life and social life, and changes in the mood. The total score of 50-59 reflects the important impact, and scores ≥60 indicate severe impact.

SECONDARY OUTCOMES:
Change from Baseline in Head Posture at 4 weeks | Baseline, 4 weeks
  Head posture is defined as the craniovertebral angle. It is the angle formed by the intersection of a horizontal line along the spinous process of C7 and the line drawn towards the ear tragus. A craniovertebral angle of <48-50° is accepted as an anterior tilt of the head.
Change from Baseline in Cervical Range of Motion at 4 weeks | Baseline, 4 weeks
  A goniometer was used to measure the cervical region's range of motion (ROM). Cervical region flexion, extension, right-left lateral flexion, and right-left rotation degrees were measured and recorded.
Change from Baseline in Temporomandibular Joint Range of Motion at 4 weeks | Baseline, 4 weeks
  For maximal mouth opening, the distance between the upper and lower incisors was measured and recorded. For protrusion, the distance between the lower and upper incisors was measured horizontally by asking the patient to bring the lower jaw forward as far as possible while the posterior teeth were in contact with each other. For right and left lateral shifts, the distance between the upper and lower incisors was measured by asking the patient to slide it to the right and left separately as much as possible.
Change from Baseline in Trigger points at 4 weeks | Baseline, 4 weeks
  While the participants were in the supine position the masseter, temporalis, pyterigoideus lateralis, pyterigoideus medialis, and digastric muscles were evaluated. In the sitting position, the sternoclavicular, suboccipital, and upper trapezius muscles were palpated, and the trigger points in these muscles and their number were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur Tuncer, Study Director — Hasan Kalyoncu University
Locations (1):
- Türkoğlu Dr. Kemal Beyazıt State Hospital, Kahramanmaraş, Turkey (Türkiye)